CLINICAL TRIAL: NCT03527732
Title: Efficacy and Safety of Ivermectin and Albendazole Co-administration in School-aged Children and Adults Infected With Trichuris Trichiura: a Multi-country Randomized Controlled Trial
Brief Title: Efficacy and Safety of IVM/ALB Co-administration
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jennifer Keiser (Other)
Collaborators: Centre Suisse de Recherches Scientifiques en Cote d'Ivoire (Other); Lao Tropical and Public Health Institute (Other Government); Public Health Laboratory of Pemba, Tanzania (Other)
Responsible Party: Sponsor-Investigator, Jennifer Keiser, Prof. Jennifer Keiser, PhD, Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2018-05-03; First posted 2018-05-17 (Actual); Results first posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2023-08

CONDITIONS: Trichuriasis
MeSH Terms: conditions — Trichuriasis | interventions — Albendazole; Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The parallel group trial will be double blinded (i.e. study participants and the trial team/researchers conducting the treatment and assessing the outcomes will be blinded) using repacked tablets including appearance-matched placebos while the dose-finding study will be single blinded (i.e. all outcome assessors except the investigators who provide the treatment and the study participants who get either active or placebo tablets matching in appearance will be blinded) due to the nature of this study (i.e. including ascending doses).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: albendazole (Placebo Comparator): 400 mg albendazole single tablet (Zentel®) and 200µg/kg using 3mg tablets of placebo at day 0 administered orally
  Interventions: Drug: Albendazole
- Arm B: albendazole and ivermectin (Experimental): 400 mg albendazole single tablet (Zentel®) and 200µg/kg using 3mg tablets of ivermectin (Stromectol®) at day 0 administered orally
  Interventions: Drug: Albendazole and Ivermectin

INTERVENTIONS:
Drug: Albendazole — Monotherapy of albendazole (400 mg)
  Other Names: Zentel®
  Arms: Arm A: albendazole
Drug: Albendazole and Ivermectin — Combination therapy of albendazole (400 mg) and ivermectin (200 µg/kg)
  Other Names: Zentel® and Stromectol®
  Arms: Arm B: albendazole and ivermectin

SUMMARY:
This study is a double-blind randomized clinical trial conducted with two settings in Africa and one in Asia, namely Côte d'Ivoire, Pemba (Zanzibar, Tanzania) and Lao PDR. This study aims at providing evidence on the efficacy and safety of co-administered albendazole and ivermectin versus albendazole monotherapy (standard of care) against whipworm (T. trichiura) infections in children and adults (6-60 years).

The efficacy of the treatment and potential extended effects on follow-up prevalence will be determined 14-21 days, 6 months and 12 months post-treatment by collecting another two stool samples. The cure rate will be calculated as the percentage of egg-positive subjects at baseline who become egg-negative after treatment.

DETAILED DESCRIPTION:
This study is a double-blind randomized clinical trial which aims at providing evidence on the efficacy and safety of co-administered albendazole and ivermectin versus albendazole monotherapy (standard of care) against T. trichiura infections in children and adults (6-60 years) in different transmission settings and geographies. Embedded in this trial a smaller dose-finding (DF) study with the goal to investigate efficacy, safety and pharmacokinetic parameters of ascending doses of ivermectin ((i) 200 µg/kg, (ii) 400 µg/kg, and (iii) 600 µg/kg) co-administered with albendazole (400 mg) in school-aged children infected with T. trichiura will take place.

The primary objective of the trial is to comparatively assess the efficacy in terms of cure rate against T. trichiura infections among school-aged children and adults from three different epidemiological settings and monitored over a 12-month period of albendazole/ivermectin combination therapy and albendazole monotherapy. A DF study will be implemented in the trial with the objective to understand the dose-dependent efficacy and pharmacokinetic profile of the co-administration of albendazole and ivermectin in school-aged children (6-12 years) with the following four oral treatment regimens: i) albendazole (400 mg) /ivermectin (200 µg/kg) combination, ii) albendazole (400 mg) /ivermectin (400 µg/kg) combination, iii) albendazole (400 mg) /ivermectin (600 µg/kg) combination, and iv) placebo.

The secondary objectives of the trial are to evaluate the safety and tolerability of the treatment regimens, compare the ERRs of the treatment regimens (combination vs. monotherapy and ascending doses of the combination) against T. trichiura, determine the CRs and ERRs of the drugs in study participants (6-60 years) infected with hookworm, A lumbricoides and S stercoralis, investigate potential extended effects on follow-up helminth prevalences (6 and 12 months post-treatment) of the two standard-dose treatment regimens (as assessed among participants with cleared infection on days 21 and 180), compare CRs based on infection status determined by novel polymerase chain reaction (PCR)-based and standard microscopic diagnosis, assess potential differences in susceptibility to the treatment regimen between the three hookworm species, Necator americanus, Ancylostoma duodenale and A. ceylanicum, as classified through the novel PCR-based diagnosis, characterize T. trichiura strains from different epidemiological settings through genotyping, evaluate potential benefits from deworming on morbidity (clinically evaluated and self-rated from questionnaire interviews) and nutritional indicators, and determine an exposure (including length of time that the drug concentration is above the minimal inhibitory concentration (MIC), Cmax, area under the curve (AUC))-response correlation of ivermectin and albendazole in school-aged children.

After obtaining informed consent from individual/parents and/or caregiver, the medical history of the participants will be assessed with a standardized questionnaire, in addition to a clinical examination carried out by the study physician before treatment. Enrollment will be based on two stool samples will be collected, if possible, on two consecutive days or otherwise within a maximum of 5 days. All stool samples will be examined with duplicated Kato-Katz thick smears by experienced laboratory technicians.

Randomization of participants into the two treatment arms will be stratified according to intensity of infection. All participants will be interviewed before treatment, 3 and 24 hours and 3 weeks after treatment about the occurrence of adverse events. Children aged 6-16 years will additionally be asked to rate their own physical functioning by replying to a pre-tested questionnaire at baseline and 6 and 12 months after treatment. The efficacy of the treatment and potential extended effects on follow-up prevalence will be determined 14-21 days, 6 months and 12 months post-treatment by collecting another two stool samples. Subjective treatment satisfaction will be assessed 3 hours, 3 weeks and 6 months after treatment to investigate relationship with treatment compliance and observed efficacy in reducing egg output and morbidity.

The primary analysis will include all participants with primary end point data (available case analysis). Supplementary, a per-protocol analysis will be conducted. CRs will be calculated as the percentage of egg-positive subjects at baseline who become egg-negative after treatment. Differences among CRs (between treatment arms and between diagnostic approaches) will be analysed by using crude and adjusted logistic regression modeling (adjustment for age, sex and weight).

Geometric and arithmetic mean egg counts will be calculated for the different treatment arms before and after treatment to assess the corresponding ERRs. Bootstrap resampling method with 5,000 replicates will be used to calculate 95% confidence intervals (CIs) for differences in ERRs.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed by either the participant him/herself (≥21 years of age) or by parents and/or caregivers for children/adolescents; and written assent by child/adolescent (aged 6-20 years).
2. Agree to comply with study procedures, including provision of two stool samples at the beginning (baseline) and on three follow-up assessments (approximately 3 weeks, 6 months, and 12 months later).
3. Aged ≥6 to <= 60 years for parallel group trial and ≥6 to <=12 years for DF study.
4. At least two slides of the quadruple Kato-Katz thick smears positive for T. trichiura and infection intensities of at least 100 EPG.

Exclusion Criteria:

1. No written informed consent by individual/parents and/or caregiver.
2. Presence of major systemic illnesses, e.g. severe anemia (below 80 g/l Hb according to WHO [28]), clinical malaria as assessed by a medical doctor (positive Plasmodium RDT and ≥38 °C ear temperature), upon initial clinical assessment.
3. History of acute or severe chronic disease (e.g. cancer, diabetes, chronic heart, liver or renal disease).
4. Recent use of anthelmintic drug (within past 4 weeks).
5. Attending other clinical trials during the study.
6. Negative or low egg count (less than 100 EPG or less than 2 out of 4 slides positive) diagnostic result for T. trichiura eggs in the stool.
7. Known allergy to study medications (i.e. albendazole and ivermectin).
8. Pregnancy or lactating in the 1st week after birth (according to WHO guidelines within LF control programs [29]).
9. Currently taking medication with known interaction (e.g. for albendazole: cimetidine, praziquantel and dexamethasone; for ivermectin: warfarin).

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1673 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Centre Suisse de Recherches Scientifiques en Côte d'Ivoire (CSRS), Abidjan, Côte d’Ivoire
- Lao Tropical and Public Health Institute, Vientiane, Laos
- Public Health Laboratory Ivo de Carneri, P.O. Box 122, Chake Chake, Pemba, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Welsche S, Schneeberger PHH, Hattendorf J, Sayasone S, Hurlimann E, Keiser J. Egg excretion patterns of soil-transmitted helminth infections in humans following albendazole-ivermectin and albendazole treatment. PLoS Negl Trop Dis. 2024 Mar 22;18(3):e0012073. doi: 10.1371/journal.pntd.0012073. eCollection 2024 Mar. PMID 38517907
- [Derived] Schneeberger PHH, Gueuning M, Welsche S, Hurlimann E, Dommann J, Haberli C, Frey JE, Sayasone S, Keiser J. Different gut microbial communities correlate with efficacy of albendazole-ivermectin against soil-transmitted helminthiases. Nat Commun. 2022 Feb 25;13(1):1063. doi: 10.1038/s41467-022-28658-1. PMID 35217670
- [Derived] Hurlimann E, Keller L, Patel C, Welsche S, Hattendorf J, Ali SM, Ame SM, Sayasone S, Coulibaly JT, Keiser J. Efficacy and safety of co-administered ivermectin and albendazole in school-aged children and adults infected with Trichuris trichiura in Cote d'Ivoire, Laos, and Pemba Island, Tanzania: a double-blind, parallel-group, phase 3, randomised controlled trial. Lancet Infect Dis. 2022 Jan;22(1):123-135. doi: 10.1016/S1473-3099(21)00421-7. Epub 2021 Nov 29. PMID 34856181
- [Derived] Keller L, Welsche S, Patel C, Sayasone S, Ali SM, Ame SM, Hattendorf J, Hurlimann E, Keiser J. Long-term outcomes of ivermectin-albendazole versus albendazole alone against soil-transmitted helminths: Results from randomized controlled trials in Lao PDR and Pemba Island, Tanzania. PLoS Negl Trop Dis. 2021 Jun 30;15(6):e0009561. doi: 10.1371/journal.pntd.0009561. eCollection 2021 Jun. PMID 34191812
- [Derived] Patel C, Hurlimann E, Keller L, Hattendorf J, Sayasone S, Ali SM, Ame SM, Coulibaly JT, Keiser J. Efficacy and safety of ivermectin and albendazole co-administration in school-aged children and adults infected with Trichuris trichiura: study protocol for a multi-country randomized controlled double-blind trial. BMC Infect Dis. 2019 Mar 18;19(1):262. doi: 10.1186/s12879-019-3882-x. PMID 30885157

RESULTS

PARTICIPANT FLOW:
Groups:
- Albendazole in Côte d'Ivoire: 400 mg albendazole single tablet (Zentel®) and placebo tablets (corresponding number to ivermectin weight-dependent dosing) at day 0 administered orally to community members aged 6-60 years in Côte d'Ivoire
- Albendazole and Ivermectin in Côte d'Ivoire: 400 mg albendazole single tablet (Zentel®) and 200µg/kg using 3mg tablets of ivermectin (Stromectol®) at day 0 administered orally to community members aged 6-60 years in Côte d'Ivoire
- Albendazole in Laos: 400 mg albendazole single tablet (Zentel®) and placebo tablets (corresponding number to ivermectin weight-dependent dosing) at day 0 administered orally to community members aged 6-60 years in Laos
- Albendazole and Ivermectin in Laos: 400 mg albendazole single tablet (Zentel®) and 200µg/kg using 3mg tablets of ivermectin (Stromectol®) at day 0 administered orally to community members aged 6-60 years in Laos
- Albendazole in Pemba Island: 400 mg albendazole single tablet (Zentel®) and placebo tablets (corresponding number to ivermectin weight-dependent dosing) at day 0 administered orally to community members aged 6-60 years in Pemba Island
- Albendazole and Ivermectin in Pemba Island: 400 mg albendazole single tablet (Zentel®) and 200µg/kg using 3mg tablets of ivermectin (Stromectol®) at day 0 administered orally to community members aged 6-60 years in Pemba Island
Period: Overall Study
Arm/Group | Albendazole in Côte d'Ivoire | Albendazole and Ivermectin in Côte d'Ivoire | Albendazole in Laos | Albendazole and Ivermectin in Laos | Albendazole in Pemba Island | Albendazole and Ivermectin in Pemba Island
Started | 256 | 255 | 274 | 275 | 305 | 308
Completed | 235 | 232 | 194 | 213 | 293 | 288
Not Completed | 21 | 23 | 80 | 62 | 12 | 20
Not completed — Lost to Follow-up | 21 | 23 | 80 | 62 | 12 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Albendazole in Côte d'Ivoire | Albendazole and Ivermectin in Côte d'Ivoire | Albendazole in Laos | Albendazole and Ivermectin in Laos | Albendazole in Pemba Island | Albendazole and Ivermectin in Pemba Island | Total
Number analyzed (Participants) | 256 | 255 | 274 | 275 | 305 | 308 | 1673
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.5 (14.1) | 16.0 (13.4) | 27.7 (17.3) | 25.9 (17.4) | 14.0 (10.5) | 13.9 (9.6) | 18.9 (15.0)
Age, Customized [Number; unit: participants]
  School-aged (6-12 years) | 171 | 168 | 92 | 113 | 191 | 184 | 919
  Youth or young people (13-24 years) | 30 | 36 | 37 | 30 | 81 | 90 | 304
  Adults (25-60 years) | 55 | 51 | 145 | 132 | 33 | 34 | 450
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 129 | 144 | 147 | 171 | 169 | 880
  Male | 136 | 126 | 130 | 128 | 134 | 139 | 793
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: kg] | 37.5 (20.1) | 37.2 (19.7) | 41.1 (14.5) | 39.7 (15.7) | 34.2 (15.5) | 34.0 (14.8) | 37.2 (16.9)
Height [Mean (Standard Deviation); unit: cm] — Population: One individual value from the Albendazole group in Laos omitted due to irrational value (479 cm).
  cm
    number analyzed (Participants) | 256 | 255 | 273 | 275 | 305 | 308 | 1672
    (all) | 136.7 (20.3) | 135.8 (19.4) | 144.3 (16.6) | 142.3 (16.7) | 137.3 (18.6) | 137.7 (18.9) | 139.0 (18.7)
T. trichiura geometric mean egg counts [Geometric Mean (Inter-Quartile Range); unit: Eggs per gram of stool] | 481 [192 to 1040] | 470 [174 to 954] | 366 [174 to 678] | 349 [168 to 618] | 467 [198 to 894] | 461 [198 to 955] | 429 [186 to 846]
T. trichiura infection intensity [Count of Participants; unit: Participants]
  Light (1-999 EPG) | 190 | 192 | 232 | 232 | 231 | 234 | 1311
  Moderate (1000-9999 EPG) | 64 | 60 | 42 | 42 | 74 | 71 | 353
  heavy (≥10 000 EPG) | 2 | 3 | 0 | 1 | 0 | 3 | 9
A. lumbricoides geometric mean egg counts [Geometric Mean (Inter-Quartile Range); unit: Eggs per gram of stool] — Population: Only A. lumbricoides co-infected participants considered.
  Eggs per gram of stool
    number analyzed (Participants) | 91 | 91 | 112 | 96 | 74 | 90 | 554
    (all) | 5499 [1020 to 24744] | 4130 [1104 to 26022] | 3991 [1161 to 18315] | 3635 [1389 to 12435] | 4515 [1938 to 11892] | 2979 [1272 to 8652] | 4036 [1284 to 15690]
A. lumbricoides infection intensity [Count of Participants; unit: Participants] — Population: Only A. lumbricoides co-infected participants considered.
  Participants
    number analyzed (Participants) | 91 | 91 | 112 | 96 | 74 | 90 | 554
    Light (1-4999 EPG) | 38 | 42 | 58 | 48 | 35 | 52 | 273
    Moderate (5000-49 999 EPG) | 40 | 39 | 47 | 44 | 38 | 37 | 245
    Heavy (≥50 000 EPG) | 13 | 10 | 7 | 4 | 1 | 1 | 36
Hookworm geometric mean egg counts [Geometric Mean (Inter-Quartile Range); unit: Eggs per gram of stool] — Population: Only hookworm co-infected participants considered.
  Eggs per gram of stool
    number analyzed (Participants) | 31 | 18 | 250 | 253 | 53 | 42 | 647
    (all) | 82 [36 to 240] | 91 [24 to 186] | 805 [390 to 2172] | 840 [348 to 2202] | 100 [36 to 294] | 80 [24 to 210] | 501 [168 to 1692]
Hookworm infection intensity [Count of Participants; unit: Participants] — Population: Only hookworm co-infected participants considered.
  Participants
    number analyzed (Participants) | 31 | 18 | 250 | 253 | 53 | 42 | 647
    Light (1-1999 EPG) | 31 | 16 | 182 | 184 | 53 | 42 | 508
    Moderate (2000-3999 EPG) | 0 | 0 | 37 | 43 | 0 | 0 | 80
    Heavy (≥4000 EPG) | 0 | 2 | 31 | 26 | 0 | 0 | 59
S. stercoralis infection [Count of Participants; unit: Participants] — Population: Baermann technique to detect S. stercoralis infection was applied only to stool samples collected in Laos; two participants (one in each group) had no S. stercoralis result.
  Participants
    number analyzed (Participants) | 0 | 0 | 273 | 274 | 0 | 0 | 547
    (all) | 0 | 0 | 29 | 30 |  |  | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants T. Trichiura Egg Negative Post-Treatment (Cured)
Description: The conversion from being egg positive pre-treatment to egg negative post-treatment, or cure rate (CR).
Time Frame: 14-21 days after treatment
Population: An analysis set of all randomized participants who provided any follow-up data was used to perform an available-case analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Albendazole in Côte d'Ivoire | Albendazole and Ivermectin in Côte d'Ivoire | Albendazole in Laos | Albendazole and Ivermectin in Laos | Albendazole in Pemba Island | Albendazole and Ivermectin in Pemba Island
Number analyzed (Participants) | 235 | 232 | 194 | 213 | 293 | 288
Participants
  Cured | 24 | 32 | 16 | 140 | 18 | 140
  Not cured | 211 | 200 | 178 | 73 | 275 | 148

2. Secondary Outcome: Number of Participants T. Trichiura Egg Negative Post-Treatment (Cured) After 6 and 12 Months Post Treatment
Description: Conversion of T. trichiura egg-positive participants at baseline who become egg-negative 6 and 12 months after treatment.
Time Frame: 6 and 12 months after treatment
Population: An analysis set of all randomized participants who provided any follow-up data at 6 or 12 months post treatment was used to perform an available-case analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Albendazole in Laos | Albendazole and Ivermectin in Laos | Albendazole in Pemba Island | Albendazole and Ivermectin in Pemba Island
Number analyzed (Participants) | 232 | 234 | 282 | 276
Participants
  Cured at 6 months | 31 | 154 | 4 | 49
  Cured at 12 months: number analyzed (Participants) | 205 | 208 | 264 | 251
  Cured at 12 months | 48 | 154 | 9 | 49

3. Secondary Outcome: Egg-reduction Rate (ERR) Against T. Trichiura
Description: Eggs per gram of stool (EPG) will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. Geometric and arithmetic mean egg counts will be calculated for the two treatment arms before and after treatment to assess the corresponding ERRs.
Time Frame: 14-21 days, 6 months and 12 months after treatment
Population: Overall number of participants analyzed corresponds to all participants that got randomized. An analysis set of all randomized participants who provided any follow-up data was used to perform an available-case analysis for each assessment time point (i.e., 14-21 days, 6 months and 12 months post-treatment).
Measure: Geometric Mean (95% Confidence Interval); unit: percent of change
Arm/Group | Albendazole in Côte d'Ivoire | Albendazole and Ivermectin in Côte d'Ivoire | Albendazole in Laos | Albendazole and Ivermectin in Laos | Albendazole in Pemba Island | Albendazole and Ivermectin in Pemba Island
Number analyzed (Participants) | 256 | 255 | 232 | 234 | 293 | 288
percent of change
  Geometric mean ERR at 14-21 days post treatment: number analyzed (Participants) | 256 | 255 | 194 | 213 | 293 | 288
  Geometric mean ERR at 14-21 days post treatment | 64 [54 to 72] | 70 [61 to 77] | 69 [61 to 75] | 99 [99 to 99] | 57 [48 to 65] | 98 [98 to 99]
  Geometric mean ERR at 6 months post treatment: number analyzed (Participants) | 0 | 0 | 232 | 234 | 282 | 276
  Geometric mean ERR at 6 months post treatment |  |  | 79.6 [73.8 to 84.3] | 99.0 [98.6 to 99.3] | 21.2 [8.1 to 33.0] | 84.9 [80.7 to 88.2]
  Geometric mean ERR at 12 months post treatmentpost treatment: number analyzed (Participants) | 0 | 0 | 205 | 208 | 264 | 251
  Geometric mean ERR at 12 months post treatmentpost treatment |  |  | 91.3 [88.5 to 93.5] | 99.6 [99.4 to 99.7] | 53.6 [45.4 to 60.9] | 92.9 [91.0 to 94.5]

4. Secondary Outcome: Number of Participants With Concomitant Soil-transmitted Helminth Infections Egg Negative Post-Treatment (Cured)
Description: Number of participants that converted from egg positive with Ascaris lumbricoides, hookworm and/or Strongyloides stercoralis infections to egg negative after 14-21 days. Number of egg-negatives at 6 and 12 months after treatment.
Time Frame: 14-21 days, 6 months and 12 months after treatment
Population: Overall number of participants include all randomized participants. To assess the number of cured 14-21 days post-treatment only randomized baseline egg positive participants with follow-up stool data were considered. For the 6 and 12 month assessment all randomized participants with at least one stool sample analyzed were considered. The number cured as assessed 14-21 days post-treatment provides a proportion that is considered the cure rate (conversion rate from positive to negative).
Measure: Count of Participants; unit: Participants
Arm/Group | Albendazole in Côte d'Ivoire | Albendazole and Ivermectin in Côte d'Ivoire | Albendazole in Laos | Albendazole and Ivermectin in Laos | Albendazole in Pemba Island | Albendazole and Ivermectin in Pemba Island
Number analyzed (Participants) | 82 | 81 | 232 | 234 | 282 | 276
Participants
  Cured from Ascaris lumbricoides at 14-21 d post treatment: number analyzed (Participants) | 82 | 81 | 77 | 70 | 70 | 86
  Cured from Ascaris lumbricoides at 14-21 d post treatment | 78 | 76 | 77 | 70 | 68 | 85
  Egg negative for Ascaris lumbricoides 6 months post treatment: number analyzed (Participants) | 0 | 0 | 232 | 234 | 282 | 276
  Egg negative for Ascaris lumbricoides 6 months post treatment |  |  | 172 | 184 | 205 | 215
  Egg negative for Ascaris lumbricoides 12 months post treatment: number analyzed (Participants) | 0 | 0 | 205 | 208 | 264 | 251
  Egg negative for Ascaris lumbricoides 12 months post treatment |  |  | 166 | 170 | 60 | 66
  Cured from hookworm 14-21 d post treatment: number analyzed (Participants) | 28 | 17 | 180 | 194 | 49 | 39
  Cured from hookworm 14-21 d post treatment | 27 | 15 | 100 | 115 | 40 | 28
  Egg negative for hookworm 6 months post treatment: number analyzed (Participants) | 0 | 0 | 232 | 234 | 282 | 276
  Egg negative for hookworm 6 months post treatment |  |  | 111 | 117 | 262 | 262
  Egg negative for hookworm 12 months post treatment: number analyzed (Participants) | 0 | 0 | 205 | 208 | 264 | 251
  Egg negative for hookworm 12 months post treatment |  |  | 126 | 146 | 250 | 231
  Cured from Strongyloides stercoralis 14-21 d post treatment: number analyzed (Participants) | 0 | 0 | 22 | 22 | 0 | 0
  Cured from Strongyloides stercoralis 14-21 d post treatment |  |  | 18 | 21 |  |

5. Secondary Outcome: Egg-reduction Rates (ERRs) Against Concomitant Soil-transmitted Helminth Infections.
Description: Percent change in geometric mean eggs per gram of stool from before to after treatment. ERRs will be calculated for Ascaris lumbricoides and hookworm infections as described in outcome 3.
Time Frame: 14-21 days, 6 months and 12 months after treatment
Population: An analysis set of all randomized participants who provided any follow-up data (14-21 days, 6 or 12 months post treatment) was used to perform an available-case analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: percent of change
Arm/Group | Albendazole in Côte d'Ivoire | Albendazole and Ivermectin in Côte d'Ivoire | Albendazole in Laos | Albendazole and Ivermectin in Laos | Albendazole in Pemba Island | Albendazole and Ivermectin in Pemba Island
Number analyzed (Participants) | 82 | 81 | 232 | 234 | 282 | 276
percent of change
  ERRs in A. lumbricoides co-infected 14-21 days post treatment: number analyzed (Participants) | 82 | 81 | 77 | 70 | 70 | 86
  ERRs in A. lumbricoides co-infected 14-21 days post treatment | 100 [100 to 100] | 100 [100 to 100] | 100 [100 to 100] | 100 [100 to 100] | 100 [100 to 100] | 100 [100 to 100]
  Extended ERRs for A. lumbricoides 6 month post treatment: number analyzed (Participants) | 0 | 0 | 232 | 234 | 282 | 276
  Extended ERRs for A. lumbricoides 6 month post treatment |  |  | 82.2 [66.1 to 90.9] | 75.8 [54.1 to 87.4] | -5.7 [-76.6 to 37.7] | 47.4 [6.1 to 69.5]
  Extended ERRs for A. lumbricoides 12 month post treatment: number analyzed (Participants) | 0 | 0 | 205 | 208 | 264 | 251
  Extended ERRs for A. lumbricoides 12 month post treatment |  |  | 87.3 [73.6 to 94.0] | 77.0 [52.3 to 89.0] | 25.0 [-36.2 to 58.6] | 48.0 [5.1 to 70.9]
  ERRs in hookworm co-infected 14-21 days post treatment: number analyzed (Participants) | 28 | 17 | 180 | 194 | 49 | 39
  ERRs in hookworm co-infected 14-21 days post treatment | 100 [100 to 100] | 99 [97 to 100] | 99 [98 to 99] | 99 [99 to 100] | 99 [97 to 100] | 97 [93 to 99]
  Extended ERRs for hookworm 6 month post treatment: number analyzed (Participants) | 0 | 0 | 232 | 234 | 282 | 276
  Extended ERRs for hookworm 6 month post treatment |  |  | 96.6 [94.9 to 97.7] | 97.7 [96.4 to 98.4] | 72.2 [56.3 to 84.1] | 73.2 [58.1 to 86.1]
  Extended ERRs for hookworm 12 month post treatment: number analyzed (Participants) | 0 | 0 | 205 | 208 | 264 | 251
  Extended ERRs for hookworm 12 month post treatment |  |  | 98.8 [98.1 to 99.2] | 99.2 [98.7 to 99.5] | 74.5 [57.5 to 87.0] | 59.2 [40.2 to 74.9]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed 3h and 24h post treatment.
Description: Adverse events were examined through standard questionnaires, graded into mild, moderate and severe (using Common Toxicity Criteria version 2.0 put forth by the Cancer Therapy Evaluation Program) and study physicians were asked to classify relatedness with drug administration in the most common expected adverse events. If causality could not be ruled out by other conditions or reasons, the adverse events were considered as possibly related.
Arm/Group | Albendazole in Côte d'Ivoire | Albendazole and Ivermectin in Côte d'Ivoire | Albendazole in Laos | Albendazole and Ivermectin in Laos | Albendazole in Pemba Island | Albendazole and Ivermectin in Pemba Island
All-Cause Mortality (participants affected / at risk) | 0/254 | 0/254 | 0/273 | 0/273 | 0/305 | 0/308
Serious Adverse Events (participants affected / at risk) | 0/254 | 0/254 | 0/273 | 0/273 | 0/305 | 0/308
Other Adverse Events (participants affected / at risk) | 83/254 | 99/254 | 77/273 | 72/273 | 28/305 | 18/308
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albendazole in Côte d'Ivoire (N=254) | Albendazole and Ivermectin in Côte d'Ivoire (N=254) | Albendazole in Laos (N=273) | Albendazole and Ivermectin in Laos (N=273) | Albendazole in Pemba Island (N=305) | Albendazole and Ivermectin in Pemba Island (N=308)
Abdominal pain (Gastrointestinal disorders) | 33 (35) | 31 (32) | 20 (22) | 10 (10) | 15 (15) | 7 (8)
Allergic reaction (Skin and subcutaneous tissue disorders) | 9 (9) | 11 (11) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — allergy-like syndromes including rash, itching and potentially also involving digestive disorders
Diarrhea (Gastrointestinal disorders) | 13 (13) | 25 (29) | 6 (6) | 3 (3) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 8 (8) | 9 (9) | 8 (8) | 0 (0) | 0 (0) — Fever was defined as body temperature of 38°C and above.
Headache (Nervous system disorders) | 26 (29) | 32 (36) | 51 (57) | 52 (63) | 8 (8) | 9 (9)
Vomiting (Gastrointestinal disorders) | 3 (3) | 10 (10) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 33 (37) | 44 (47) | 2 (2) | 7 (7) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (10) | 11 (11) | 4 (4) | 8 (8) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/32/NCT03527732/Prot_SAP_000.pdf